CLINICAL TRIAL: NCT00134563
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Design Study to Evaluate the Efficacy and Safety of Teriflunomide in Reducing the Frequency of Relapses and Delaying the Accumulation of Physical Disability in Subjects With Multiple Sclerosis With Relapses
Brief Title: Study of Teriflunomide in Reducing the Frequency of Relapses and Accumulation of Disability in Patients With Multiple Sclerosis
Acronym: TEMSO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC6049; 2004-000555-42 (EudraCT Number); HMR1726D/3001 (Other: HMR)
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing Remitting; Secondary Progressive; Progressive Relapsing
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Teriflunomide 7 mg (Experimental): Teriflunomide 7 mg once daily for 108 weeks
  Interventions: Drug: Teriflunomide
- Teriflunomide 14 mg (Experimental): Teriflunomide 14 mg once daily for 108 weeks
  Interventions: Drug: Teriflunomide
- Placebo (Placebo Comparator): Placebo (for teriflunomide) once daily for 108 weeks
  Interventions: Drug: Placebo (for teriflunomide)

INTERVENTIONS:
Drug: Teriflunomide — Film-coated tablet
  Oral administration
  Other Names: HMR1726
  Arms: Teriflunomide 14 mg; Teriflunomide 7 mg
Drug: Placebo (for teriflunomide) — Film-coated tablet
  Oral administration
  Arms: Placebo

SUMMARY:
The primary objective was to determine the effect of teriflunomide on the frequency of relapses in patients with relapsing multiple sclerosis (MS).

Secondary objectives were:

* to evaluate the effect of teriflunomide on the accumulation of disability as measured by Expanded Disability Status Scale [EDSS], the burden of disease as measured by Magnetic Resonance Imaging [MRI] and patient-reported fatigue;
* to evaluate the safety and tolerability of teriflunomide.

DETAILED DESCRIPTION:
The study period per participant was approximatively 128 weeks broken down as follows:

* Screening period up to 4 weeks,
* 108-week double-blind treatment period (approximatively 2 years)*,
* 16-week post-treatment elimination follow-up period.

'*' Participants successfully completing the week 108 visit were offered the opportunity to enter the optional long-term extension study LTS6050 - NCT00803049.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis [MS] subject who was ambulatory (EDSS of ≤ 5.5)
* Exhibiting a relapsing clinical course, with or without progression (relapsing remitting, secondary progressive or progressive relapsing);
* Meeting McDonald's criteria for MS diagnosis;
* Experienced at least 1 relapse over the 1 year preceding the trial or at least 2 relapses over the 2 years preceding the trial;
* No relapse onset in the preceding 60 days prior to randomization;
* Clinically stable during the 30 days prior to randomization, without adrenocorticotrophic hormone [ACTH] or systemic steroid treatment.

Exclusion Criteria:

* Clinically relevant cardiovascular, hepatic, neurological, endocrine or other major systemic disease;
* Significantly impaired bone marrow function;
* Pregnant or nursing woman;
* Alcohol or drug abuse;
* Use of cladribine, mitoxantrone, or other immunosuppressant agents such as azathioprine, cyclophosphamide, cyclosporin, methotrexate or mycophenolate before enrollment;
* Any known condition or circumstance that would prevent in the investigator's opinion compliance or completion of the study;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1088 (Actual)
Dates: Start 2004-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Connor, MD, Principal Investigator — St. Michael's Hospital (Toronto, Canada)
Locations (21):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis Austria, Vienna, Austria
- sanofi-aventis, Canada, Laval, Canada
- Sanofi-Aventis, Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- sanofi-aventis Denmark, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- sanofi-aventis Finland, Helsinki, Finland
- sanofi-aventis France, Paris, France
- Sanofi-Aventis Deutschland GmbH, Berlin, Germany
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Lysaker, Norway
- sanofi-aventis Poland, Warsaw, Poland
- Sanofi-Aventis, Porto Salvo, Portugal
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Bromma, Sweden
- Sanofi-Aventis Switzerland, Geneva, Switzerland
- sanofi-aventis Turkey, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Kiev, Ukraine
- sanofi-aventis UK, Guildford, Surrey, United Kingdom

REFERENCES:
- [Result] O'Connor P, Wolinsky JS, Confavreux C, Comi G, Kappos L, Olsson TP, Benzerdjeb H, Truffinet P, Wang L, Miller A, Freedman MS; TEMSO Trial Group. Randomized trial of oral teriflunomide for relapsing multiple sclerosis. N Engl J Med. 2011 Oct 6;365(14):1293-303. doi: 10.1056/NEJMoa1014656. PMID 21991951
- [Derived] Sprenger T, Kappos L, Sormani MP, Miller AE, Poole EM, Cavalier S, Wuerfel J. Effects of teriflunomide treatment on cognitive performance and brain volume in patients with relapsing multiple sclerosis: Post hoc analysis of the TEMSO core and extension studies. Mult Scler. 2022 Oct;28(11):1719-1728. doi: 10.1177/13524585221089534. Epub 2022 Apr 29. PMID 35485424
- [Derived] Comi G, Freedman MS, Meca-Lallana JE, Vermersch P, Kim BJ, Parajeles A, Edwards KR, Gold R, Korideck H, Chavin J, Poole EM, Coyle PK. Prior treatment status: impact on the efficacy and safety of teriflunomide in multiple sclerosis. BMC Neurol. 2020 Oct 6;20(1):364. doi: 10.1186/s12883-020-01937-4. PMID 33023488
- [Derived] Radue EW, Sprenger T, Gaetano L, Mueller-Lenke N, Cavalier S, Thangavelu K, Panzara MA, Donaldson JE, Woodward FM, Wuerfel J, Wolinsky JS, Kappos L. Teriflunomide slows BVL in relapsing MS: A reanalysis of the TEMSO MRI data set using SIENA. Neurol Neuroimmunol Neuroinflamm. 2017 Aug 9;4(5):e390. doi: 10.1212/NXI.0000000000000390. eCollection 2017 Sep. PMID 28828394
- [Derived] Sormani MP, Truffinet P, Thangavelu K, Rufi P, Simonson C, De Stefano N. Predicting long-term disability outcomes in patients with MS treated with teriflunomide in TEMSO. Neurol Neuroimmunol Neuroinflamm. 2017 Jun 28;4(5):e379. doi: 10.1212/NXI.0000000000000379. eCollection 2017 Sep. PMID 28680917
- [Derived] Freedman MS, Wolinsky JS, Comi G, Kappos L, Olsson TP, Miller AE, Thangavelu K, Benamor M, Truffinet P, O'Connor PW; TEMSO and TOWER Study Groups. The efficacy of teriflunomide in patients who received prior disease-modifying treatments: Subgroup analyses of the teriflunomide phase 3 TEMSO and TOWER studies. Mult Scler. 2018 Apr;24(4):535-539. doi: 10.1177/1352458517695468. Epub 2017 Mar 17. PMID 28304217
- [Derived] Miller AE, O'Connor P, Wolinsky JS, Confavreux C, Kappos L, Olsson TP, Truffinet P, Wang L, D'Castro L, Comi G, Freedman MS; Teriflunomide Multiple Sclerosis Trial Group. Pre-specified subgroup analyses of a placebo-controlled phase III trial (TEMSO) of oral teriflunomide in relapsing multiple sclerosis. Mult Scler. 2012 Nov;18(11):1625-32. doi: 10.1177/1352458512450354. Epub 2012 Jun 21. PMID 22723573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment initiated in September 2004 was completed in February 2008.
  A total of 1338 patients were screened at 127 sites in 21 countries.
Pre-assignment Details: Randomization was stratified by country and baseline disability (Expanded Disability Status Scale [EDSS] score ≤3.5 or >3.5).
  Assignment to groups was done centrally using an Interactive Voice Response System (IVRS] in a 1:1:1 ratio after confirmation of the selection criteria.
  1088 participants were randomized.
Period: Overall Study
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Started | 363 (Randomized) | 366 (Randomized) | 359 (Randomized)
Treated | 363 (Two participants received doses of Teriflunomide 7 mg, one participant doses of Teriflunomide 14 mg) | 365 | 358 (one participant received doses of Teriflunomide 7 mg)
Completed | 259 (completed treatment period) | 274 (completed treatment period) | 263 (completed treatment period)
Not Completed | 104 | 92 | 96
Not completed — Not treated due to protocol violation | 0 | 1 | 1
Not completed — Adverse Event | 29 | 37 | 38
Not completed — Lack of Efficacy | 24 | 14 | 17
Not completed — Protocol Violation | 3 | 2 | 5
Not completed — Lost to Follow-up | 4 | 0 | 2
Not completed — progressive disease | 11 | 4 | 2
Not completed — did not wish to continue | 33 | 32 | 26
Not completed — Reason other than above | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg | Total
Number analyzed (Participants) | 363 | 365 | 358 | 1086
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics of the population included in analyses
  years | 38.4 (9.0) | 37.5 (9.0) | 37.8 (8.2) | 37.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 254 | 254 | 783
  Male | 88 | 111 | 104 | 303
Region of enrollment [Number; unit: participants] — America: Canada, Chile, and United States;
  Eastern Europe: Czech Republic, Estonia, Poland, Russia and Ukraine;
  Western Europe: Austria, Denmark, Finland, France, Germany, Italy, Netherlands, Norway, Portugal, Sweden, Switzerland, Turkey, and United Kingdom;
  participants
    America | 82 | 83 | 80 | 245
    Eastern Europe | 114 | 116 | 108 | 338
    Western Europe | 167 | 166 | 170 | 503
Time since first diagnosis of multiple sclerosis (MS) [Mean (Standard Deviation); unit: Years] — The information was missing for one participant in the Teriflunomide 7 mg group.
  Years | 5.13 (5.59) | 5.29 (5.36) | 5.59 (5.44) | 5.33 (5.48)
Number of MS relapses [Median (Full Range); unit: MS relapses]
  Within the past year | 1 [0 to 6] | 1 [0 to 6] | 1 [0 to 4] | 1 [0 to 6]
  Within the past 2 years | 2 [1 to 7] | 2 [1 to 12] | 2 [1 to 9] | 2 [1 to 12]
Time since most recent MS relapse onset [Mean (Standard Deviation); unit: months] | 6.28 (3.62) | 6.29 (3.29) | 6.50 (3.71) | 6.35 (3.54)
MS subtype [Number; unit: participants]
  Relapsing Remitting | 329 | 332 | 332 | 993
  Secondary Progressive | 22 | 17 | 12 | 51
  Progressive Relapsing | 12 | 16 | 14 | 42
MS medication in the past 2 years [Number; unit: participants]
  Yes | 90 | 102 | 102 | 294
  No | 273 | 263 | 256 | 792
Baseline EDSS total score [Number; unit: participants] — EDSS is an ordinal scale in half-point increments that qualifies disability in patients with MS. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation.
  EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  participants
    ≤ 3.5 | 281 | 280 | 276 | 837
    > 3.5 | 82 | 85 | 82 | 249

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate [ARR]: Poisson Regression Estimates
Description: ARR is obtained from the total number of confirmed relapses that occured during the treatment period divided by the sum of the treatment durations.
  Each episode of relapse - appearance, or worsening of a clinical symptom that was stable for at least 30 days, that persisted for a minimum of 24 hours in the absence of fever - was to be confirmed by an increase in EDSS score or Functional System scores.
  To account for the different treatment durations among participants, a Poisson regression model with robust error variance was used (total number of confirmed relapses as response variable; log-transformed treatment duration as "offset" variable; treatment group, region of enrollment and baseline EDSS stratum as covariates).
Time Frame: 108 weeks
Population: All randomized and treated participants; Participants were included in the treatment group to which they were originally assigned (intent-to-treat analysis).
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 363 | 365 | 358
relapses per year | 0.539 [0.466 to 0.623] | 0.370 [0.318 to 0.432] | 0.369 [0.308 to 0.441]
Statistical Analysis 1: Comparison: Placebo vs Teriflunomide 14 mg; Null hypothesis: * H1: No difference between Teriflunomide 14 mg and placebo * H2: No difference between Teriflunomide 7 mg and placebo The study was sized to detect a 25% relative risk reduction with teriflunomide in the 2-year relapse rate at a significance level of 0.050 with a power ≥95% anticipating a potential 20% 2-year dropout rate; Test type: Superiority or Other; p = 0.0005, Regression, Poisson — Step down approach used to adjust for multiplicity: * H1 tested first * H2 tested only if the comparison H1 was statistically significant A priori threshold for statistical significance for both comparisons ≤0.05; Relative risk reduction (%) = 31.5 — Relative risk reduction with Teriflunomide 14 mg compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Teriflunomide 7 mg; Test type: Superiority or Other; p = 0.0002, Regression, Poisson — [p-value comment as in outcome 1, analysis 1]; Relative Risk Reduction (%) = 31.2 — Relative risk reduction with Teriflunomide 7 mg compared to placebo

2. Secondary Outcome: Time to 12-week Sustained Disability Progression: Kaplan-Meier Estimates of the Rate of Disability Progression at Timepoints
Description: 12-week sustained disability progression was defined as an increase from baseline of at least 1-point in EDSS score (at least 0.5-point for participants with baseline EDSS score >5.5) that persisted for at least 12 weeks.
  Probability of disability progression at 24, 48 and 108 weeks was estimated using Kaplan-Meier method on the time to disability progression defined as the time from randomization to first EDSS increase. Participants free of disability progression (no disability progression observed on treatment) were censored at the date of the last on-treatment EDSS evaluation.
  Kaplan-Meier method consists in computing probabilities of non occurrence of event at any observed time of event and multiplying successive probabilities for time ≤t by any earlier computed probabilities to estimate the probability of being event-free for the amount of time t. Probability of event at time t is 1 minus the probability of being event-free for the amount of time t.
Time Frame: 108 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 363 | 365 | 358
percent probability
  Probability of disability progression at 24 weeks | 8.6 [5.7 to 11.6] | 5.8 [3.3 to 8.3] | 6.2 [3.6 to 8.8]
  Probability of disability progression at 48 weeks | 16.0 [12.1 to 20.0] | 13.1 [9.4 to 16.7] | 11.3 [7.9 to 14.8]
  Probability of disability progression at 108 weeks | 27.3 [22.3 to 32.3] | 21.7 [17.1 to 26.3] | 20.2 [15.6 to 24.7]
Statistical Analysis 1: Comparison: Placebo vs Teriflunomide 14 mg; Null hypothesis: * H1: No difference between Teriflunomide 14 mg and placebo * H2: No difference between Teriflunomide 7 mg and placebo The study was also sized to detect a 37% hazard rate reduction of an assumed disability progression hazard rate of 0.1783 in the placebo group and 0.1116 in the teriflunomide group by the end of 2 years with a power of 80% anticipating a potential 20% 2-year dropout rate; Test type: Superiority or Other; p = 0.0279, Log Rank — Step down approach: * H1 tested only if both comparisons on the primary outcome measure were statistically significant * H2 tested only if the comparison H1 was statistically significant A priori threshold for statistical significance ≤0.05; Two-sided Log-rank test stratified by region of enrollment and baseline EDSS stratum; Hazard ratio reduction (%) = 29.8 — Relative risk reduction with Teriflunomide 14 mg compared to placebo (estimated from a Cox proportional hazard model with treatment arm, region of enrollment and baseline EDSS stratum as covariates)
Statistical Analysis 2: Comparison: Placebo vs Teriflunomide 7 mg; Test type: Superiority or Other; p = 0.0835, Log Rank — [p-value comment as in outcome 2, analysis 1]; Two-sided Log-rank test stratified by region of enrollment and baseline EDSS stratum; Hazard ratio reduction (%) = 23.7 — Relative risk reduction with Teriflunomide 7 mg compared to placebo (estimated from a Cox proportional hazard model with treatment arm, region of enrollment and baseline EDSS stratum as covariates)

3. Secondary Outcome: Cerebral Magnetic Resonance Imaging [MRI] Assessment: Change From Baseline in Total Lesion Volume (Burden of Disease)
Description: Total lesion volume is the sum of the total volume of all T2-lesions and the total volume all T1-hypointense post-gadolinium lesions measured through T2/proton density scan analysis and gadolinium-enhanced T1 scan analysis.
Time Frame: baseline (before randomization) and 108 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mililiters (mL)
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 363 | 365 | 358
mililiters (mL)
  Change in total lesion volume | 2.208 (7.002) | 1.308 (6.799) | 0.723 (7.591)
  - Change in T1-hypointense lesion component | 0.533 (1.063) | 0.499 (1.154) | 0.331 (1.012)
  - Change in T2-lesion component | 1.674 (6.473) | 0.810 (6.181) | 0.392 (6.901)
Statistical Analysis 1: Comparison: Placebo vs Teriflunomide 14 mg; Mixed-effect model with repeated measures [MMRM] on cubic root transformed total lesion volume data (treatment group, region of enrollment, baseline EDSS stratum, visit, treatment-by-visit interaction, baseline value (cubic root transformed) and baseline-by-visit interaction); Test type: Superiority or Other; p = 0.0003, t-test, 2 sided — A priori threshold for statistical significance ≤0.05 No adjustment for multiple comparisons; 2-sided t-test on baseline adjusted least-square means
Statistical Analysis 2: Comparison: Placebo vs Teriflunomide 7 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0317, t-test, 2 sided — A priori threshold for statistical significance ≤0.05 No adjustment for multiple comparisons; 2-sided t-test on baseline adjusted least-square means

4. Other Pre Specified Outcome: Cerebral MRI Assessment: Number of Gd-enhancing T1-lesions Per Scan (Poisson Regression Estimates)
Description: Number of Gd-enhancing T1-lesions per scan is obtained from the total number of Gd-enhancing T1-lesions observed during the study divided by the total number of scans performed during the study.
  To account for the different number of scans among participants, a Poisson regression model with robust error variance was used (total number of Gd-enhancing T1-lesions as response variable; log-transformed number of scans as "offset" variable; treatment group, region of enrollment, baseline EDSS stratum and baseline number of Gd-enhancing T1-lesions as covariates).
Time Frame: 108 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 346 | 350 | 340
lesions per scan | 1.331 [1.059 to 1.673] | 0.570 [0.434 to 0.748] | 0.261 [0.167 to 0.407]

5. Other Pre Specified Outcome: Cerebral MRI Assessment: Volume of Gd-enhancing T1-lesions Per Scan
Description: Total volume of Gd-enhancing T1-lesions per scan is obtained from the sum of the volumes of Gd-enhancing T1-lesions observed during the study divided by the total number of scans performed during the study.
Time Frame: 108 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mililiters (mL)
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 346 | 350 | 340
mililiters (mL) | 0.102 (0.329) | 0.059 (0.247) | 0.025 (0.079)

6. Secondary Outcome: Changes From Baseline in Fatigue Impact Scale [FIS] Total Score
Description: FIS is a subject-reported scale that qualifies the impact of fatigue on daily life in patients with MS. It consists of 40 statements that measure fatigue in three areas; physical, cognitive, and social.
  FIS total score ranges from 0 (no problem) to 160 (extreme problem).
  Least-square means were estimated using a Mixed-effect model with repeated measures [MMRM] on FIS total score data (treatment group, region of enrollment, baseline EDSS stratum, visit, treatment-by-visit interaction, baseline value, and baseline-by-visit interaction as factors).
Time Frame: baseline (before randomization) and 108 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Number analyzed (Participants) | 363 | 365 | 358
units on a scale | 4.300 (1.670) [-98 to 99] | 2.343 (1.641) [-114 to 96] | 3.804 (1.670) [-86 to 95]
Statistical Analysis 1: Comparison: Placebo vs Teriflunomide 14 mg; Test type: Superiority or Other; p = 0.8271, t-test, 2 sided — A priori threshold for statistical significance ≤0.05 No adjustment for multiple comparisons; 2-sided t-test on baseline adjusted least-square means
Statistical Analysis 2: Comparison: Placebo vs Teriflunomide 7 mg; Test type: Superiority or Other; p = 0.3861, t-test, 2 sided — A priori threshold for statistical significance ≤0.05 No adjustment for multiple comparisons; 2-sided t-test on baseline adjusted least-square means

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected regardless of seriousness or relationship to the drug, spanning from signature of the Informed Consent Form up to the last visit.
Description: The analysis was performed on the exposed population and included all AE that developed or worsened from first study drug intake up to 112 days after last intake or up to first intake in the extension study, whichever came first (124 weeks max).
  Participants who received incorrect treatment were included considering the incorrect treatment.
Arm/Group | Placebo | Teriflunomide 7 mg | Teriflunomide 14 mg
Serious Adverse Events (participants affected / at risk) | 46/360 | 52/368 | 57/358
Other Adverse Events (participants affected / at risk) | 259/360 | 271/368 | 265/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=360) | Teriflunomide 7 mg (N=368) | Teriflunomide 14 mg (N=358)
Appendicitis (Infections and infestations) | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 3
Renal abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 2 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Psychosomatic disease (Psychiatric disorders) | 0 | 1 | 0
Somatoform disorder (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0
Glossopharyngeal neuralgia (Nervous system disorders) | 1 | 0 | 0
Hypertonia (Nervous system disorders) | 1 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 3 | 0 | 3
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 4
Intestinal functional disorder (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 6 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 2
Post abortion haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 2 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 5 | 5
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Nuclear magnetic resonance imaging abdominal abnormal (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 2 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus operation (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=360) | Teriflunomide 7 mg (N=368) | Teriflunomide 14 mg (N=358)
Bronchitis (Infections and infestations) | 22 | 18 | 29
Gastroenteritis (Infections and infestations) | 15 | 22 | 20
Influenza (Infections and infestations) | 35 | 34 | 43
Nasopharyngitis (Infections and infestations) | 98 | 94 | 93
Sinusitis (Infections and infestations) | 16 | 15 | 23
Upper respiratory tract infection (Infections and infestations) | 25 | 34 | 32
Urinary tract infection (Infections and infestations) | 35 | 27 | 36
Depression (Psychiatric disorders) | 27 | 26 | 33
Insomnia (Psychiatric disorders) | 23 | 20 | 15
Dizziness (Nervous system disorders) | 16 | 22 | 17
Headache (Nervous system disorders) | 64 | 81 | 67
Hypoaesthesia (Nervous system disorders) | 30 | 18 | 20
Paraesthesia (Nervous system disorders) | 30 | 34 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 15 | 19
Abdominal pain (Gastrointestinal disorders) | 24 | 17 | 21
Abdominal pain upper (Gastrointestinal disorders) | 15 | 19 | 20
Diarrhoea (Gastrointestinal disorders) | 32 | 54 | 64
Nausea (Gastrointestinal disorders) | 26 | 32 | 49
Vomiting (Gastrointestinal disorders) | 14 | 15 | 18
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 38 | 47
Rash (Skin and subcutaneous tissue disorders) | 15 | 14 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 30 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 46 | 39 | 40
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 | 16 | 13
Muscular weakness (Musculoskeletal and connective tissue disorders) | 23 | 15 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 47 | 26 | 33
Fatigue (General disorders) | 51 | 47 | 52
Alanine aminotransferase increased (Investigations) | 21 | 41 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results of the work performed pursuant to this protocol. Prior to publication, the investigator provides the sponsor with the manuscript for review and comment at least 45 days in advance of its submission for publication.

The sponsor can require the investigator to withhold publication an additional 90 days to allow for filing a patent application or taking such other measures as sponsor deems appropriate to establish and preserve its proprietary rights.